CLINICAL TRIAL: NCT05112913
Title: A Double-blind, Randomized Clinical Trial to Evaluate the Lot-to-lot Consistency, Immunogenicity and Safety of an Inactivated SARS-CoV-2 Vaccine (CoronaVac）Between Different Workshops for Prevention of COVID-19 in Healthy Children Aged 3-17 Years
Brief Title: Lot-to-lot Consistency of an Inactivated SARS-CoV-2 Vaccine Between Different Workshops in Healthy Children Aged 3-17 Years
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sinovac Research and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-nCOV-MA4006-SN
Record Dates: First submitted 2021-11-08; First posted 2021-11-09 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — SARS-CoV-2 inactivated vaccines; sinovac COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Inactivated SARS-CoV-2 vaccine Lot 1 of the workshop 2 (Experimental): 360 Participants aged 3-17 years(including 52 children aged 3-5 years,154 children aged 6-11 years and 154 adolescents aged 12-17 years) will receive Inactivated SARS-CoV-2 vaccine Lot 1 of the workshop 2 according to 0,28-day immunization schedule.
  Interventions: Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell) Lot 1 of the workshop 2
- Inactivated SARS-CoV-2 vaccine Lot 2 of the workshop 2 (Experimental): 360 Participants aged 3-17 years(including 52 children aged 3-5 years,154 children aged 6-11 years and 154 adolescents aged 12-17 years) will receive Inactivated SARS-CoV-2 vaccine Lot 2 of the workshop 2 according to 0,28-day immunization schedule.
  Interventions: Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell) Lot 2 of the workshop 2
- Inactivated SARS-CoV-2 vaccine Lot 3 of the workshop 2 (Experimental): 360 Participants aged 3-17 years(including 52 children aged 3-5 years,154 children aged 6-11 years and 154 adolescents aged 12-17 years) will receive Inactivated SARS-CoV-2 vaccine Lot 3 of the workshop 2 according to 0,28-day immunization schedule.
  Interventions: Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell) Lot 3 of the workshop 2
- Inactivated SARS-CoV-2 vaccine Lot 1 of the workshop 3 (Experimental): 360 Participants aged 3-17 years(including 52 children aged 3-5 years,154 children aged 6-11 years and 154 adolescents aged 12-17 years) will receive Inactivated SARS-CoV-2 vaccine Lot 1 of the workshop 3 according to 0,28-day immunization schedule.
  Interventions: Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell) Lot 1 of the workshop 3
- Inactivated SARS-CoV-2 vaccine Lot 2 of the workshop 3 (Experimental): 360 Participants aged 3-17 years(including 52 children aged 3-5 years,154 children aged 6-11 years and 154 adolescents aged 12-17 years) will receive Inactivated SARS-CoV-2 vaccine Lot 2 of the workshop 3 according to 0,28-day immunization schedule.
  Interventions: Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell) Lot 2 of the workshop 3
- Inactivated SARS-CoV-2 vaccine Lot 3 of the workshop 3 (Experimental): 360 Participants aged 3-17 years(including 52 children aged 3-5 years,154 children aged 6-11 years and 154 adolescents aged 12-17 years) will receive Inactivated SARS-CoV-2 vaccine Lot 3 of the workshop 3 according to 0,28-day immunization schedule.
  Interventions: Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell) Lot 3 of the workshop 3
- Inactivated SARS-CoV-2 vaccine Lot 1 of the workshop 1 (Active Comparator): 360 Participants aged 3-17 years(including 52 children aged 3-5 years,154 children aged 6-11 years and 154 adolescents aged 12-17 years) will receive Inactivated SARS-CoV-2 vaccine Lot 1 of the workshop 1 according to 0,28-day immunization schedule.
  Interventions: Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell) Lot 1 of the workshop 1

INTERVENTIONS:
Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell) Lot 1 of the workshop 2 — 600SU inactivated virus in 0.5 mL of aluminium hydroxide solution per injection
  Other Names: CoronaVac
  Arms: Inactivated SARS-CoV-2 vaccine Lot 1 of the workshop 2
Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell) Lot 2 of the workshop 2 — 600SU inactivated virus in 0.5 mL of aluminium hydroxide solution per injection
  Other Names: CoronaVac
  Arms: Inactivated SARS-CoV-2 vaccine Lot 2 of the workshop 2
Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell) Lot 3 of the workshop 2 — 600SU inactivated virus in 0.5 mL of aluminium hydroxide solution per injection
  Other Names: CoronaVac
  Arms: Inactivated SARS-CoV-2 vaccine Lot 3 of the workshop 2
Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell) Lot 1 of the workshop 3 — 600SU inactivated virus in 0.5 mL of aluminium hydroxide solution per injection
  Other Names: CoronaVac
  Arms: Inactivated SARS-CoV-2 vaccine Lot 1 of the workshop 3
Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell) Lot 2 of the workshop 3 — 600SU inactivated virus in 0.5 mL of aluminium hydroxide solution per injection
  Other Names: CoronaVac
  Arms: Inactivated SARS-CoV-2 vaccine Lot 2 of the workshop 3
Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell) Lot 3 of the workshop 3 — 600SU inactivated virus in 0.5 mL of aluminium hydroxide solution per injection
  Other Names: CoronaVac
  Arms: Inactivated SARS-CoV-2 vaccine Lot 3 of the workshop 3
Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell) Lot 1 of the workshop 1 — 600SU inactivated virus in 0.5 mL of aluminium hydroxide solution per injection
  Other Names: CoronaVac
  Arms: Inactivated SARS-CoV-2 vaccine Lot 1 of the workshop 1

SUMMARY:
This study is a double-blind, randomized phase Ⅳ clinical trial of the inactivated SARS-CoV-2 vaccine (CoronaVac)manufactured by Sinovac Research & Development Co., Ltd. The purpose of this study is to evaluate the lot-to-lot consistency ,immunogenicity and safety of COVID-19 vaccine between the commercialized scale in workshop 2 and 3 and the commercialized scale in workshop 1 in healthy children aged 3-17 years.

DETAILED DESCRIPTION:
This study is a double-blind, randomized phase Ⅳ clinical trial in healthy children aged 3-17 years to evaluate the lot-to-lot consistency, immunogenicity and safety of the commercial-scale CoronaVac in healthy children aged 3-17 years .The experimental vaccine was manufactured by Sinovac Research & Development Co.,Ltd. A total of 2520 healthy subjects aged 3 to 17 years old will be enrolled.The subjects will be randomly divided into 7 groups of 360 participants per group with an equal probability to received 7 batches of commercial-scale vaccine.All subjects received two doses of vaccine on day 0 and day 28.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 3-17;
* The subjects and/or guardians can understand and voluntarily sign the informed consent form (For subjects aged 8-17 years, both subjects and guardians need to sign the informed consent form)
* Proven legal identity.

Exclusion Criteria:

* History of SARS-CoV-2 infection;
* History of receiving COVID-19 vaccine;
* History of asthma, history of allergy to the vaccine or vaccine components, or serious adverse reactions to the vaccine, such as urticaria, dyspnea,and angioedema;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;
* Autoimmune disease (Systemic lupus erythematosus)or immunodeficiency / immunosuppression(HIV,history after organ transplantation)
* Severe chronic diseases, severe cardiovascular diseases, hypertension and diabetes that cannot be controlled by drugs, liver or kidney diseases, malignant tumors, etc.;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Thyroid disease or history of thyroidectomy,absence of spleen, functional absence of spleen, absence of spleen due to any condition or splenectomy;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* Receipt of blood products within in the past 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Onset of various acute or chronic diseases within 7 days prior to the study;
* Axillary temperature >37.0°C;
* The subjects participated in other clinical trials during the follow-up period, or will be planned within 3 months;
* Already pregnant (including a positive urine pregnancy test) or are breastfeeding, planning to get pregnant within 2 months;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2520 (Estimated)
Dates: Start 2021-07-27 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titer(GMT) of neutralizing antibody to live SARS-CoV-2 | 28 days after the full immunization
  Geometric mean titer(GMT) of neutralizing antibody to live SARS-CoV-2 28 days after the full immunization of each lot of COVID-19 vaccine

SECONDARY OUTCOMES:
Geometric mean increase (GMI) of the neutralizing antibody to live SARS-CoV-2 | 28 days after the full immunization
  Geometric mean increase (GMI) of the neutralizing antibody to live SARS-CoV-2 28 days after the full immunization of each lot of COVID-19 vaccine
Seroconversion rate of the neutralizing antibody to live SARS-CoV-2 | 28 days after the full immunization
  Seroconversion rate of the neutralizing antibody to live SARS-CoV-2 28 days after the full immunization of each lot of COVID-19 vaccine
Seropositivity rate of the neutralizing antibody to live SARS-CoV-2 | 28 days after the full immunization
  Seropositivity rate of the neutralizing antibody to live SARS-CoV-2 28 days after the full immunization of each lot of COVID-19 vaccine
Incidence of adverse reactions 0-7 days after vaccination | 0-7 days after vaccination
  The incidence of adverse reactions of each lot of COVID-19 vaccine 0-7 days after vaccination
Incidence of adverse reactions 0-28 days after vaccination | 0-28 days after vaccination
  The incidence of adverse reactions of each lot of COVID-19 vaccine 0-28 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Weijun Hu, Master, Principal Investigator — Shanxi Provincial Center for Disease Prevention and Control
Locations (1):
- Yaliang county Center for Disease Control and Prevention, Xi’an, Shanxi, China